CLINICAL TRIAL: NCT00274014
Title: Effects of Inhaled Tiotropium Bromide on Severity of Airflow Obstruction During Long-term Treatment in Patients With Moderately Severe Copd. Impact on Severity and Incidence of Exacerbations.
Brief Title: Measure of the Long Term Influence of SPIRIVA® in Acute Respiratory Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.214
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
The objectives of this study were to evaluate the effect of a one-year treatment with inhaled tiotropium bromide 18 mcg once daily on lung function, incidence and severity of exacerbations in patients with chronic obstructive pulmonary disease (COPD).

The secondary purpose was to explore possible relationships between lung function changes and occurrence of COPD exacerbations and to try to characterize these exacerbations.

DETAILED DESCRIPTION:
This was a multicentre, randomised, double blind, parallel group, placebo-controlled, one year study. It was designed to determine the effect of inhaled tiotropium treatment on airflow obstruction (PEFR), incidence and severity of exacerbations in patients with COPD.

Following an initial 3-week screening period qualifying patients were randomized to either tiotropium or placebo at Visit 2. Patients returned to the clinic at weeks 6 (Visit 3), 12 (Visit 4), 24 (Visit 5), 36 (Visit 6), 48 (Visit 7) and at Week 50 for the conclusion of the trial (Visit 8). The patients received treatment daily for 48 weeks (336 days).

PEFR, as well as use of rescue medication and respiratory condition, were self-assessed by patients and recorded every morning on a graphical diary card every morning. The graphical presentation of these data was supposed to help investigators to detect exacerbations occurring between two consecutive visits.

Details on hospitalizations due to COPD exacerbations were recorded in a special hospitalization booklet.

Study Hypothesis:

The objectives of this study were to evaluate the effect of a one-year treatment with inhaled tiotropium bromide 18 mcg once daily on lung function, incidence and severity of exacerbations in patients with chronic obstructive pulmonary disease (COPD).

The secondary purpose was to explore possible relationships between lung function changes and occurrence of COPD exacerbations and to try to characterize these exacerbations.

Comparison(s):

Tiotropium 18 mcg once daily vs Placebo

ELIGIBILITY:
* Diagnosis of COPD according to the European Respiratory Society (ERS) (R95-3225) and matching the following criteria:

  * Stable moderate to severe airway obstruction
  * Baseline 30 % < FEV1 < 65 % of European Community of Coal and Steel (ECCS) predicted values (R94-1408).
  * Baseline FEV1/SVC< 70 %.
* Smoking history > 10 pack-years (p.y.). A p.y. was defined as the equivalent of smoking
* One pack of cigarettes per day for one year.
* History of exacerbation in the past year.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2000-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10

PRIMARY OUTCOMES:
morning peak expiratory flow rate (PEFR) | 50 weeks

SECONDARY OUTCOMES:
incidence, severity and duration of exacerbations | 50 weeks
number of patients with one or more exacerbation | 50 weeks
rate of PEFR drops | 50 weeks
number of lost working days | 50 weeks
number of days of hospitalisation | 50 weeks
use of rescue medications, type and duration | 50 weeks
bacterial and viral characterisation of severe exacerbations | 50 weeks
spirometric evaluation (FEV1, FVC, SVC, MEF25-75 ) and optional measurements (IC) | 50 weeks
plethysmography (RV, TLC) (optional) | 50 weeks
Adverse events, physical examination | 50 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI France S.A.S.
Locations (53):
- France (53):
  - Clinique Saint Sauveur, Angers
  - Boehringer Ingelheim Investigational Site, Annecy
  - Clinique la Casamance, Aubagne
  - Boehringer Ingelheim Investigational Site, Avrillé
  - Hôpital, Bois-Guillaume
  - GPL, Caluire-et-Cuire
  - Boehringer Ingelheim Investigational Site, Châlons-en-Champagne
  - CH Cholet, Cholet
  - Boehringer Ingelheim Investigational Site, Cholet
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Clinique des Cèdres, Cornebarrieu
  - Clinique Saint Vincent, Épernay
  - Centre Hospitalier Auban Moet, Épernay
  - Boehringer Ingelheim Investigational Site, Le Blanc-Mesnil
  - Boehringer Ingelheim Investigational Site, Le Petit-Quevilly
  - Hôpital Calmette, Lille
  - Boehringer Ingelheim Investigational Site, Lyon
  - CH Lyon Sud, Lyon
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Louis Pradel, Lyon
  - Boehringer Ingelheim Investigational Site, Marseille
  - Hôpital Ambroise Paré, Marseille
  - Hôpital Nord, Marseille
  - CHG, Martigues
  - Boehringer Ingelheim Investigational Site, Metz
  - Hôpital N.D. bon Secours, Metz
  - Service des maladies respiratoires, Montpellier
  - Centre Hospitalier Universitaire Arnaud de Villeneuve, Montpellier
  - Polyclinique Les Fleurs, Ollioules
  - Hôpital Hôtel Dieu, Paris
  - Hôpital St Antoine, Paris
  - CTAR, Paris
  - Fondation Saint Joseph, Paris
  - Hôpital Cochin, Paris
  - Hôpital Bichat-Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - Groupe Médical Saint Rémi, Reims
  - Hôpital Charles Nicolle, Rouen
  - CHILTERN, Rueil-Malmaison
  - CHD Félix Guyon, Saint Denis de La Réunion
  - Nouvelle Clinique Union et Vaurais, Saint-Jean
  - Centre Hospitalier Sud-Réunion, Saint-Pierre
  - Boehringer Ingelheim Investigational Site, Salon-de-Provence
  - Boehringer Ingelheim Investigational Site, Saumur
  - Boehringer Ingelheim Investigational Site, Sélestat
  - Boehringer Ingelheim Investigational Site, Strasbourg
  - Hôpital Hautepierre, Strasbourg
  - CHU Purpan, Toulouse
  - Cabinet de Pneumologie, Toulouse
  - Cabinet Médical, Toulouse
  - Clinique Saint Jean Lanquedoc, Toulouse
  - CHU Rangueil, Toulouse
  - Centre Hospitalier, Villefranche-sur-Saône